CLINICAL TRIAL: NCT06597175
Title: A Multi-center, Open-label, Single Arm, Prospective Pivotal Medical Device Clinical Trial to Evaluate Efficacy and Safety of Study Device (ORIGO) That Provides Numerical Data by Measuring the Composition Within Breast Tissue Using Diffusion Optical Spectroscopy Imaging Technology to Assist in the Differential Diagnosis of Breast Tumors in Patients With Breast Lesions
Brief Title: Evaluating Investigational Medical Device for Breast Tumor Diagnosis Using Diffusion Optical Spectroscopy
Acronym: ORIGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Olive Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ORIGO_E23-01
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Breast Tumor; Mammary Carcinoma, Human
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Device: ORIGO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device: ORIGO (Experimental)
  Interventions: Device: ORIGO

INTERVENTIONS:
Device: ORIGO — The device measurement is first performed on the breast area with the lesion, followed by the measurement of the corresponding area in the contralateral breast for comparison.

SUMMARY:
This is a multicenter, pivotal clinical trial to evaluate the safety and efficacy of a diagnostic device used to assist in the differentiation of breast tumors in patients with breast lesions detected by ultrasound alone or by both ultrasound and mammography.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 19 years or older
* ACR BI-RADS Category 3-5 (5th edition, 2023 update)

Exclusion Criteria:

* Pregnant, potentially pregnant, or currently breastfeeding
* Calcifications detected on mammography but do not have corresponding lesions identified on ultrasound
* Biopsy performed on the same breast within 7 days prior to the date of informed consent
* Significant trauma or scarring at the measurement site, or those suffering from mastitis.
* Breast implants, electronic medical devices such as pacemakers, or with a space left in the breast cavity due to implant removal
* History of phototoxic reactions or light sensitivity

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Concordance | Through study completion, an average of 6 months
  Concordance between biopsy results (Gold standard) and the device test results for breast lesions in subjects

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Seoul
  - Yongin Severance Hospital, Yongin-si

IPD SHARING:
Plan to Share IPD: No